CLINICAL TRIAL: NCT00450892
Title: A Phase I-II Study of Lapatinib and Docetaxel as Neoadjuvant Treatment for HER-2 Positive Locally Advanced/Inflammatory or Large Operable Breast Cancer
Brief Title: Phase I/II Study of Neoadjuvant Lapatinib in Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-10054; EORTC-10054; GSK-EORTC-10054; 2006-000864-94 (EudraCT Number)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: inflammatory breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Docetaxel; Trastuzumab; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- arm 1 (Other)
  Interventions: Drug: docetaxel+lapatinib
- arm 2 (Other)
  Interventions: Drug: docetaxel + trastuzumab
- arm 3 (Experimental)
  Interventions: Drug: docetaxel + trastuzumab + lapatinib

INTERVENTIONS:
Drug: docetaxel+lapatinib — 3 cycles of docetaxel (100 mg/m²) + lapatinib (1000 mg/d) followed by 3 cycles of FEC
  Arms: arm 1
Drug: docetaxel + trastuzumab — 3 cycles of docetaxel (100 mg/m²) + trastuzumab weekly schedule followed by 3 cycles of FEC 100
  Arms: arm 2
Drug: docetaxel + trastuzumab + lapatinib — 3 cycles of docetaxel (100 mg/m²) + trastuzumab weekly schedule
  +lapatinib (1000 mg/d) followed by 3 cycles of FEC 100
  Arms: arm 3

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, fluorouracil, epirubicin, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving these treatments before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving trastuzumab after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This randomized phase I/II trial is studying the side effects and best dose of docetaxel and lapatinib when given with or without combination chemotherapy and to see how well they work in treating women with locally advanced, inflammatory, or resectable breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of neoadjuvant therapy comprising docetaxel and lapatinib ditosylate before or after fluorouracil, epirubicin hydrochloride, and cyclophosphamide (FEC chemotherapy) in patients with HER2-positive locally advanced, inflammatory, or large resectable breast cancer. (Phase I)
* Determine the safety of this regimen in these patients. (Phase I)
* Determine the pathological complete response rate in patients treated with neoadjuvant docetaxel and lapatinib ditosylate followed by FEC chemotherapy, and with neoadjuvant docetaxel and trastuzumab (Herceptin®) followed by FEC chemotherapy. (Phase II)

Secondary

* Determine the biological activity (i.e., changes in apoptosis and proliferation markers [PTEN mutation and function, pAkt, mTOR, and associated proteins]) of neoadjuvant docetaxel and lapatinib ditosylate in these patients. (Phase I)
* Determine adverse events or biological modifications. (Phase I)
* Determine the tolerability of these regimens in these patients. (Phase II)
* Determine the clinical activity of these regimens. (Phase II)
* Identify genes that may predict response in patients treated with docetaxel and lapatinib ditosylate. (Phase II)

OUTLINE: This is a multicenter, open-label, phase I dose-escalation study of docetaxel and lapatinib ditosylate followed by a randomized phase II study. Patients enrolled in the phase II portion of the study are stratified by institution and disease status (locally advanced disease vs large operable tumor).

* Phase I (completed as of 5/26/2010): Patients receive docetaxel IV over 1 hour on day 1 and oral lapatinib ditosylate once daily on days 1-21. Treatment repeats every 3 weeks for 4 courses. Two additional courses may be given at the discretion of the physician.

  * Cohorts of 3-6 patients receive escalating doses of docetaxel and lapatinib ditosylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT).
* Phase I bridge step (completed as of 5/26/2010): Patients receive FEC chemotherapy comprising fluorouracil IV over 15 minutes, epirubicin hydrochloride IV over 60 minutes, and cyclophosphamide IV over 60 minutes on day 1. Treatment repeats every 3 weeks for 3 courses. Patients also receive docetaxel and lapatinib ditosylate as in phase I at the MTD for up to 3 courses.

  * Cohorts of 3-6 patients receive de-escalating doses of docetaxel and lapatinib ditosylate in combination with FEC chemotherapy until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT.
* Phase II: Patients are randomized to 1 of 3 treatment arms.

  * Arm I: Patients receive docetaxel and lapatinib ditosylate at the MTD as in the bridge step of phase I followed by FEC chemotherapy.
  * Arm II: Patients receive docetaxel IV over 60 minutes and trastuzumab (Herceptin®) IV over 30-90 minutes on days 1, 8, and 15. Patients then receive FEC chemotherapy as in the bridge step of phase I. Treatment with docetaxel and trastuzumab repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.
  * Arm III: Patients receive docetaxel IV over 60 minutes, lapatinib ditosylate at the MTD as in the bridge step of phase I, and trastuzumab (Herceptin®) IV over 30-90 minutes on days 1, 8, and 15. Patients then receive FEC chemotherapy as in the bridge step of phase I. Treatment with docetaxel, lapatinib ditosylate, and trastuzumab repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

All patients then undergo surgery to remove the tumor. Patients may then receive trastuzumab every 3 weeks for 1 year.

Blood samples are collected at baseline and periodically during study for pharmacokinetic studies. Patients also undergo tumor biopsies at baseline and periodically during study for laboratory studies. Blood and tissue samples are analyzed by quantitative reverse transcriptase polymerase chain reaction for biomarker profiling (HER1-3, Akt 1-3, mTOR, RICTOR, RAPTOR, CCND1, p21, survivin, PTEN), immunohistochemistry, fluorescent in situ hybridization (TopoII, HER2), and proteomics.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for the phase II.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer meeting the following criteria:

  * Phase I

    * Locally advanced or inflammatory disease, or specified subgroup of large operable disease for whom neoadjuvant chemotherapy is appropriate, defined as any 1 of the following:

      * Clinical stage T4a-d, any N (inflammatory breast carcinoma: tumor mass, breast enlargement, oedema and warmth of the skin are often present but not mandatory for the diagnosis)
      * Any clinical T, N2 or N3 (ipsilateral supraclavicular nodes)
      * cT3cN0,1 any estrogen receptor (ER)
      * cT2cN1 any ER
      * cT2cN0 ER negative
    * Presence of bilateral breast cancer is allowed
    * No bone, liver, or other extensive metastases

      * Minimal lung, skin, or nodal metastases may be allowed at the discretion of the investigator (phase I only)
  * Phase II

    * Locally advanced or inflammatory breast cancer, defined as any 1 of the following:

      * Clinical T4a-d, any N (inflammatory breast carcinoma: tumor mass, breast enlargement, oedema and warmth of the skin are often present but not mandatory for the diagnosis)
      * Any clinical T, N2 or N3 (ipsilateral supraclavicular nodes)
      * And M0
    * Bilateral breast cancer is allowed provided only 1 side is HER2-positive
    * Any large resectable T2 or T3 breast cancers, M0
* HER2-positive disease by immunohistochemistry, fluorescent in situ hybridization, and/or chromogenic in situ hybridization
* No CNS involvement
* Two frozen trucuts for every core biopsy indicated by the translational research study
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive or negative tumor

PATIENT CHARACTERISTICS:

* Female
* WHO performance status 0-2
* Hemoglobin > 10.0 g/dL
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT < 3 times ULN
* Creatinine < 1.5 times ULN
* No other malignancies within the past 3 years except basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix (phase II)
* LVEF normal by MUGA or ECHO
* ECG normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception 2 weeks prior to, during, and for 1 month after completion of study treatment
* No current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease not requiring therapy as per investigator assessment)
* No serious cardiac illness or medical condition within the past 6 months including, but not limited to, any of the following:

  * History of documented congestive heart failure
  * High-risk uncontrolled arrhythmias
  * Angina pectoris requiring antianginal medication
  * Clinically significant valvular heart disease
  * Evidence of transmural infarction on ECG
  * Poorly controlled hypertension, defined as systolic blood pressure (BP) > 180 mm Hg or diastolic BP > 100 mm Hg
* Able to swallow and retain oral medication
* Accessible for repeat dosing and follow up
* No concurrent grapefruit juice
* No active or uncontrolled infection
* No other serious illness
* No malabsorption syndrome
* No other medical condition (i.e., history of chronic alcohol abuse, hepatitis, HIV, and/or cirrhosis)
* No psychological, familial, sociological, or geographical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

* No prior therapy for any cancer, including chemotherapy, radiotherapy, or hormonal therapy for breast cancer (phase I)
* No prior epidermal growth factor receptor- or HER2-targeted therapy or antibody therapy (phase I)
* More than 10 days since prior and no concurrent CYP3A4 inducers or inhibitors
* More than 14 days since prior and no concurrent herbal infusions or dietary supplements
* No antacids 1 hour before or after lapatinib ditosylate administration
* No other concurrent investigational therapy or anticancer therapy
* No concurrent prophylactic antibiotics

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Phase I part: Dose limiting toxicity during cycle 1 | during study
Phase II: Pathological complete response rate | end of study

SECONDARY OUTCOMES:
Phase I: Changes in apoptosis and proliferation markers. | end of Phase I
Phase II: Tolerability, clinical/radiological response rates, breast conserving surgery, pharmacodynamics data | end of study

CONTACTS AND LOCATIONS:
Overall Officials: David Cameron, MD, Study Chair — Edinburgh Cancer Centre at Western General Hospital; Herve Bonnefoi, MD, Study Chair — Institut Bergonié
Locations (15):
- Belgium (2):
  - C.H.U. Sart-Tilman, Liège
  - Clinique Sainte Elisabeth, Namur
- France (9):
  - Institut Bergonie, Bordeaux
  - Institut Bergonié, Bordeaux
  - CHRU de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - CRLC Val D'Aurelle, Montpellier
  - Centre Henri Becquerel, Rouen
  - Hopital Rene Huguenin - Institut Curie, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut Gustave Roussy, Villejuif
- The Institute Of Oncology, Ljubljana, Slovenia
- Switzerland (2):
  - Hôpitaux universitaires de Genève - HUG - site de Cluse-Roseraie, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- Western General Hospital, Edinburgh, United Kingdom

REFERENCES:
- [Result] Bonnefoi H, Jacot W, Saghatchian M, Moldovan C, Venat-Bouvet L, Zaman K, Matos E, Petit T, Bodmer A, Quenel-Tueux N, Chakiba C, Vuylsteke P, Jerusalem G, Brain E, Tredan O, Messina CG, Slaets L, Cameron D. Neoadjuvant treatment with docetaxel plus lapatinib, trastuzumab, or both followed by an anthracycline-based chemotherapy in HER2-positive breast cancer: results of the randomised phase II EORTC 10054 study. Ann Oncol. 2015 Feb;26(2):325-32. doi: 10.1093/annonc/mdu551. Epub 2014 Dec 1. PMID 25467016
- [Result] Bonnefoi H, Zaman K, Debled M, Fiche M, Fournier M, Nobahar M, Pierga JY, Koch KM, Bartlett J, Zimmer A, Marreaud S, Bogaerts J, Cameron D. An European Organisation for Research and Treatment of Cancer phase I study of lapatinib and docetaxel as neoadjuvant treatment for human epidermal growth factor receptor 2 (HER2) positive locally-advanced/inflammatory or large operable breast cancer. Eur J Cancer. 2013 Jan;49(2):281-9. doi: 10.1016/j.ejca.2012.08.006. Epub 2012 Sep 18. PMID 22999386